CLINICAL TRIAL: NCT04515212
Title: In-Field Detection of Acute Intracranial Hemorrhage Requiring Urgent, Life-Saving Treatment in Severe Traumatic Brain Injury (TBI) Patients
Brief Title: In-Field Detection of Intracranial Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Pro00104100
Record Dates: First submitted 2020-08-13; First posted 2020-08-17 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Volunteers (Active Comparator)
  Interventions: Other: Optic Nerve Ultrasounds
- Traumatic Brain Injury Patients (Experimental)
  Interventions: Other: Optic Nerve Ultrasounds

INTERVENTIONS:
Other: Optic Nerve Ultrasounds — Patients will have up to four ultrasounds of the optic nerve.

SUMMARY:
This is a research study to develop a noninvasive test using ultrasound to determine when urgent, life-saving treatment is needed for those with severe traumatic brain injuries.

ELIGIBILITY:
Healthy Volunteer Inclusion Criteria:

* Adults 18 or older
* Able to provide legally effective consent

Healthy Volunteer Exclusion Criteria:

* Intracranial disease, neurologic symptoms, or eye pathology

Patient Inclusion Criteria:

* Adults age 18 or older
* Confirmed or suspected severe traumatic brain injury
* Able to provide legally effective consent

Patient Exclusion Criteria:

* Significant bilateral ocular trauma

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2024-02-07 (Actual); Study Completion 2024-02-10 (Actual)

PRIMARY OUTCOMES:
Optic nerve sheath diameter | Approximately 10 minutes at the time of ultrasounds
  Develop software that will automatically measure optic nerve sheath diameter by analyzing the radio frequency data from an ultrasound probe intervention from those that do not, we will measure the optic nerve sheath diameter manually in the cross-sectional images.

CONTACTS AND LOCATIONS:
Overall Officials: Sean Montgomery, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-02-01): https://cdn.clinicaltrials.gov/large-docs/12/NCT04515212/ICF_000.pdf